CLINICAL TRIAL: NCT06115733
Title: A Single-arm, Single-center, Prospective Phase I/II Study of Fuquinitinib Combined With Capecitabine First-line Maintenance in the Treatment of Metastatic Colorectal Cancer
Brief Title: Study of Fuquinitinib Combined With Capecitabine First-line Maintenance in the Treatment of Metastatic Colorectal Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Qi Li, Oncology department chief physician, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-125
Record Dates: First submitted 2023-10-30; First posted 2023-11-03 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-10

CONDITIONS: Colorectal Carcinoma
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Capecitabine combined with fuquitinib (Experimental): Phase Ⅰb dose exploration trial of fuquinitinib combined with capecitabine (n=6-9) :
  1. Capecitabine: 1000 mg/m² orally, twice a day on days 1-21 of each cycle, 28 days for one treatment cycle.
  2. Fuquinitinib: 1 to 21 days per cycle, orally, once a day, 28 days for a treatment cycle. There are two dose gradients of fuquintinib: 2mg/d, and the initial dose of 3mg/d is 2mg/d. According to the 3+3 dose climbing principle, dose exploration is carried out in the order of 2mg/d→3mg/d, The recommended dose of fuquinitinib combined with capecitabine, as determined in phase I b, continued to enroll 47 patients in the dose-expansion phase trial until the patient became intolerant of toxicity or disease progression.
  Interventions: Drug: Fruquintinib、Capecitabine Tablets

INTERVENTIONS:
Drug: Fruquintinib、Capecitabine Tablets — Phase Ⅰb dose exploration trial of fuquinitinib combined with capecitabine (n=6-9) :
  3) Capecitabine: 1000 mg/m² orally, twice a day on days 1-21 of each cycle, 28 days for one treatment cycle.
  4) Fuquinitinib: 1 to 21 days per cycle, orally, once a day, 28 days for a treatment cycle. There are two dose gradients of fuquintinib: 2mg/d, and the initial dose of 3mg/d is 2mg/d. According to the 3+3 dose climbing principle, dose exploration is carried out in the order of 2mg/d→3mg/d, as follows:
  Phase II: Dose extension trial (n=47) :
  The recommended dose of fuquinitinib combined with capecitabine, as determined in phase I b, continued to enroll 47 patients in the dose-expansion phase trial until the patient became intolerant of toxicity or disease progression.

SUMMARY:
This is a single-arm, single-center, prospective phase I/II study that received standard first-line chemotherapy (FOLFOX,FOLFIRI,XELOX, FOLFOXIRI± targeted therapy). If the first-line chemotherapy regimen is a 2-week regimen, patients need to undergo ≥8 cycles of standard chemotherapy. If the first-line chemotherapy regimen is a 3-week regimen, maintenance therapy is required for patients with unresectable advanced metastatic colorectal cancer who have reached CR,PR,SD (RECIST 1.1) after standard chemotherapy after ≥4 cycles.

The eligible patients were screened for maintenance treatment. Maintenance therapy research is divided into the following two phases:

Phase IIB fuquinitinib combined capecitabine dose exploration trial (n=6-9) : Phase II: Dose extension trial (n=47) : 47 patients were continued to be enrolled in the dose extension phase trial according to the recommended dose of fuquinitinib combined with capecitabine established in phase iB, and were treated until toxicity became intolerable or disease progression.

ELIGIBILITY:
Inclusion Criteria:

* 1. Have fully understood the study and voluntarily signed the informed consent;

  2. Age 18-75 years old (including 18 and 75 years old);

  3. The patient must have histologically/cytologically proven advanced metastatic colorectal cancer;

  4. Received standard first-line chemotherapy (FOLFOX,FOLFIRI,XELOX, FOLFOXIRI± targeted therapy). If the first-line chemotherapy regimen is a 2-week regimen, patients need to undergo ≥8 cycles of standard chemotherapy. If the first-line chemotherapy regimen is a 3-week regimen, patients need to undergo ≥4 cycles of standard chemotherapy. Patients with unresectable advanced metastatic colorectal cancer who achieved CR,PR,SD (RECIST 1.1) after standard chemotherapy.

  5. Must have at least one evaluable lesion (RECIST 1.1);

  6. At least one lesion is located outside the irradiation area if prior radiotherapy has been performed;

  7.ECOG physical condition 0-1 score;

  8. Expected survival ≥12 weeks;

  9. The functions of vital organs meet the following requirements (the use of any blood components and cell growth factors is not allowed within *14 days before enrollment) :
* Absolute neutrophil count ≥1.5×109/L;
* Platelets ≥100×109/L;
* Hemoglobin ≥9g/dL;
* Serum albumin ≥3g/dL;
* Bilirubin ≤1.5 times ULN;
* ALT and AST ≤2.5 times ULN;
* Serum creatinine ≤1.5 ULN;

Fertile male or female patients volunteered to use effective contraceptive methods, such as double barrier methods, condoms, oral or injectable contraceptives, and Iuds, during the study period and within 6 months of the last study medication. All female patients will be considered fertile unless they have undergone natural menopause, artificial menopause, or sterilization (such as hysterectomy, bilateral adnexectomy, or irradiation of radioactive ovaries).

Exclusion Criteria:

* Received fuquinitinib treatment before enrollment;

  2. Participated in other domestic unapproved or unmarketed drug clinical trials and accepted the corresponding experimental drug treatment within 4 weeks before enrollment;

  3. Received TACE treatment within 6 weeks before enrollment;

  4. Received any surgery or invasive treatment or operation (except intravenous catheterization, puncture drainage, etc.) within 4 weeks before enrollment;

  5. International Standardized Ratio (INR) > 1.5 or partially activated prothrombin time (APTT) > 1.5×ULN;

  6. The investigator identified clinically significant electrolyte abnormalities;

  7. The patient currently has hypertension that cannot be controlled by drugs, as follows: systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg;

  8. The patient currently has poorly controlled diabetes (fasting glucose concentration ≥CTCAE level 2 after formal treatment);

  9. The patient has any current disease or condition that affects drug absorption, or the patient cannot take fuquintinib orally;

  10. The patient currently has gastrointestinal diseases such as active gastric and duodenal ulcers, ulcerative colitis, or active bleeding from unresectosed tumors, or other conditions determined by researchers that may cause gastrointestinal bleeding or perforation;

  11. Patients with evidence or history of significant bleeding tendency within 3 months prior to enrollment (bleeding within 3 months > 30 mL, hematemesis, stool, stool blood), hemoptysis (within 4 weeks > 5 mL of fresh blood) or had a thromboembolic event (including stroke events and/or transient ischemic attacks) within 12 months;

  12. Clinically significant cardiovascular disease, including but not limited to acute myocardial infarction, severe/unstable angina pectoris, or coronary artery bypass grafting within 6 months prior to enrollment; New York Heart Association (NYHA) Grades for Congestive Heart Failure > Level 2; Ventricular arrhythmias requiring medical treatment; LVEF (Left ventricular Ejection Fraction) < 50%;

  13. Have had other malignancies within the past 5 years, except basal cell or squamous cell carcinoma of the skin after radical surgery, or carcinoma in situ of the cervix;

  14. Active or uncontrolled severe infection (≥CTCAE v5.0 grade 2 infection);

  15. Known human immunodeficiency virus (HIV) infection; Known history of clinically significant liver disease, including viral hepatitis [Known hepatitis B virus (HBV) carriers must rule out active HBV infection, i.e., positive HBV DNA (>1×104 copies /mL or > 2000 IU/ml); known hepatitis C virus infection (HCV) and HCV RNA positive (>1×103 copies /mL), or other hepatitis, cirrhosis];

  16. The patient has current central nervous system (CNS) metastases or previous brain metastases;

  17. Unmitigated toxicity higher than CTCAE v5.0 grade 1 due to any previous anticancer therapy, excluding alopecia, lymphocytopenia, and oxaliplatin grade ≤2 neurotoxicity;

  18. Women who are pregnant (positive pregnancy test before medication) or breastfeeding;

  19. Received blood transfusion therapy, blood products and hematopoietic factors, such as albumin and granulocyte colony-stimulating factor (G-CSF), within 14 days before enrollment;

  20. Target lesions received brachytherapy (particle implantation) within 60 days before enrollment;

  21. Any other medical condition, a clinically significant metabolic abnormality, physical abnormality, or laboratory abnormality that, in the investigator's judgment, reasonably suspects the patient to have a medical condition or condition that is not suitable for the use of the investigational drug (such as the presence of epileptic seizures requiring treatment), or that would affect the interpretation of the study results, or would place the patient at high risk.

  22.Urine routine indicated urinary protein ≥2+, and 24-hour urinary protein volume > 1.0g.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2023-12-28 (Estimated); Primary Completion 2026-12-15 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
RP2D | RP2D is defined as approximately 4 months from the date of enrollment to the end of the study or the date of first recorded progress or the date of death from any cause, whichever comes first
  Recommended dose for Phase II study
PFS | PFS is defined as approximately 12 months from the date of enrollment until the date of first recorded progress or the date of death from any cause, whichever comes first
  Progression-Free Survival

SECONDARY OUTCOMES:
ORR | From date of enrollment until the end of treatment or the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
  Objective Response Rate
OS | OS From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36months
  overall survival
DCR | From date of enrollment until the end of treatment or the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
  Disease control rate

IPD SHARING:
Plan to Share IPD: No